CLINICAL TRIAL: NCT05772182
Title: Non-invasive Tool to Assess Electrophysiological Mechanisms in Cardiac Arrhythmias (SAVE-COR)
Brief Title: Non-invasive Tool to Assess Electrophysiological Mechanisms in Cardiac Arrhythmias
Acronym: SAVE-COR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corify Care S.L. (Industry)
Collaborators: Hospital General Universitario Gregorio Marañon (Other); Hospital Clinic of Barcelona (Other); Hospital Universitario La Fe (Other)
Responsible Party: Sponsor
Other Study IDs: SAVE-COR
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Cardiac Arrhythmia
Keywords: Non-invasive; Electrocardiographic imaging (ECGI)
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Groups/Cohorts: Patients undergoing intervention for arrhythmia (electrophysiologic study and/or intracardiac device implantation) with clinical indication
  Interventions: Device: ACORYS MAPPING SYSTEM

INTERVENTIONS:
Device: ACORYS MAPPING SYSTEM — Diagnostic Test: ECG-Imaging
  Diagnostic Test: Standard 12-lead ECG
  Diagnostic Test: Endocardial mapping and/or pacing

SUMMARY:
Noninvasive evaluation of the electrical status of the heart is based on the standard ECG but remains suboptimal due to difficulties with arrhythmia characterization and location. Electrocardiographic Imaging (ECGI) provides maps of cardiac electrical excitation in relation to the anatomy of the heart using an extensive number of electrodes from the body surface. The applicant will develop a systematic evaluation of the ECGI as a tool to detect cardiac regions of interest in cardiac arrhythmias.

DETAILED DESCRIPTION:
The specific aim of this multicenter observational study is to evaluate the precision of non-invasive cardiac mapping system ECGI using multipolar intracardiac recordings as the gold standard. We will develop a non-invasive ECGi and intracardiac recordings in patients undergoing electrophysiology studies and/or intracardiac devices implantation to correlate the position of the regions of interest at predefined anatomy sites in patients with different organized arrhythmias. The long-term outcome of the electrophysiological characterization using ECGI will be also evaluated. Finally, the cost-efficiency of ECGI system as a support tool in cardiac arrhythmias diagnosis will be assessed.

Objectives: to perform a systematic evaluation of the ECGI with recordings using multipolar intracardiac recordings as the gold standard. Secondly, the study will also validate the ability of the ECGI recordings to increase the precision of the standard ECG interpretation by an expert.

ELIGIBILITY:
Inclusion Criteria:

* Indication for an invasive electroanatomic study and/or intracardiac device implantation.
* Having obtained and signed the informed consent for study participation.
* Ability to stand, to be able to obtain the 3D torso reconstruction necessary for the ECGI system.

Exclusion Criteria:

* <18 years old
* Inability to perform an endocardial catheterization and/or device implantation.
* Physical or mental disability to understand and accept the informed consent.
* Inability to stand to obtain the 3D torso reconstruction.
* active coronary ischemia or decompensated heart failure
* Intracardiac clot on trans-esophageal echocardiography
* Pregnancy.
* Disorganized arrhythmias (i.e. atrial fibrillation, polymorphic ventricular tachycardia).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patient's population will include those with an indication for an invasive electroanatomic study and/or intracardiac device implantation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of ECGI for detecting cardiac region of interest | 1 year
  Accuracy of the ECGI non-invasive cardiac mapping system for detecting cardiac regions of interest in cardiac arrhythmias through direct confrontation with invasive endocardial contact measures.

SECONDARY OUTCOMES:
Correlation of ECGI with an expert's interpretation of the standard ECG | 1 year
  Correlation of ECGI with an expert's interpretation of the standard ECG in terms of identifying a cardiac region of interest in an arrhythmia.
ECGI's ability to accurately predict the success of ablation procedures and recurrence | 1 year
  Degree of concordance of the electrophysiological characterization obtained by ECGI with the success of ablation procedures and recurrence.
Cost-effectiveness rate of the ECGI | 1 year
  Cost-effectiveness rate of the ECGI as a support tool in the diagnosis of cardiac arrhythmias.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No